CLINICAL TRIAL: NCT06713694
Title: The Effectiveness of Cognitive Behavioral Therapy on Anxiety, Depression, and Stigma Among Chinese Patients With Inflammatory Bowel Disease Across Diverse Cultural Identities:Protocol for a Pilot Randomised Controlled Trial
Brief Title: The Impact of Culture in Cognitive Behavior Therapy (CBT) for Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Zhen (Other)
Responsible Party: Sponsor-Investigator, Wang Zhen, Clinical Reaserch Nurse, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ZJSRRSH202479337
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Disease (IBD); Cognitive Behavior Therapy
Keywords: inflammatory bowel disease; cognitive behavior therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be divided into high and low groups based on the results of the Chinese Confucian coping Thinking Scale assessment. After completion of the first baseline assessment, patients will be randomly assigned to the experimental or waiting-list control condition.Randomization will be stratified by gender, disease type and will be conducted by an off-site statistician not involved in patient recruitment or assessment, using random allocation software.Participants assigned to the experimental condition will start treatment as soon as possible (maximum within 6 weeks). The second, mid-treatment assessment will take place four weeks following start of treatment and the third assessment one month following completion of treatment. Following the first baseline assessment, participants assigned to the waiting-list control condition will wait 3.5 months, then they will be asked to complete a follow-up assessment after waiting/baseline before they are treated with CBT.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CBT (Experimental)
  Interventions: Other: cognitive-behavioral therapy
- CBT-II (Experimental)
  Interventions: Other: cognitive-behavioral therapy
- Wait-list (Other)
  Interventions: Other: Wait first, then cognitive-behavioral therapy
- Wait-list-II (Other)
  Interventions: Other: Wait first, then cognitive-behavioral therapy

INTERVENTIONS:
Other: cognitive-behavioral therapy — The treatment will consist of eight weekly sessions, each lasting one hour. The first session will focus on the rationale of cognitive behavioral therapy, i.e. the influence of (irrational or dysfunctional) cognitions and attitudes on (restrictive) feelings and behaviors. Additionally, goal setting will be initiated. Since patients may have a wide diversity of psychiatric problems (i.e. PTSD, anxiety disorders and depression), the treatment manual will encompass five optional modules for the therapist that focus on each of these disorders (i.e. exposure based for anxiety and PTSD, behavioral activation for depression). The subsequent sessions (2-6) will target teaching the patient to identify and challenge dysfunctional cognitions and attitudes related to IBD. Each session will address specific illness-related cognitions. If possible, dysfunctional cognitions and attitudes will be replaced by helpful cognitions and attitudes.
  Arms: CBT; CBT-II
Other: Wait first, then cognitive-behavioral therapy — participants assigned to the waiting-list control condition will wait 3.5 months before they are treated with CBT. This period corresponds to the duration of the CBT intervention and follow-up assessment of the experimental group. After this 3.5 month waiting period the participants in the waiting-list control condition will be asked to complete a follow-up after waiting/baseline before CBT assessment before starting treatment.
  Arms: Wait-list; Wait-list-II

SUMMARY:
Introduction Inflammatory bowel disease (IBD), which includes Crohn's disease and ulcerative colitis, is a chronic condition that affects the gastrointestinal tract and has a significant impact on patients' quality of life (QoL) and mental health(Barberio, Zamani et al. 2021). Cognitive behavioral therapy (CBT) has been recognized as a potential therapeutic approach to address the psychological comorbidities associated with IBD(Seaton, Hudson et al. 2024). However, the effectiveness of CBT in IBD is not solely a clinical issue but is also intertwined with cultural factors that can influence treatment outcomes(Naeem 2019).

The effectiveness of CBT in IBD is not solely a clinical issue but is also intertwined with cultural factors that can influence treatment outcomes . This has implications for the delivery of CBT in IBD care, as cultural beliefs and values can affect help-seeking behaviors and responses to treatment. Cultural factors are integral to the successful implementation of CBT in IBD care(Hinton and Patel 2017, Naeem, Sajid et al. 2023). Further research is needed to understand how cultural adaptations can enhance the efficacy of CBT for IBD patients from diverse backgrounds. It is essential to consider cultural nuances in the development and delivery of CBT to ensure that it is both effective and acceptable to patients with IBD across different cultures.

Objective: To identify gaps in the current understanding of the role of culture in CBT for IBD, including the variety of cultural contexts and IBD populations studied . To provide insights that can guide clinical practice in offering culturally competent CBT to IBD patients and inform policy decisions regarding mental health services for diverse populations with IBD .

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age with diagnosed IBD.
2. Age: 18 years and older.
3. residing in China, able to verbally communicate and read in Chinese, with access to the internet to ensure participation in the online intervention.
4. Able to commit to attend the 6weekly sessions of 1 hours' duration.
5. No change in antidepressant medication (dose or type) within 3 months of trial onset.

Exclusion Criteria:

1. Individuals scheduled for major surgery in the next 3 months.
2. Current psychological treatment.
3. Individuals with severe schizophrenia/psychotic disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
mood | From enrollment to the end of treatment at 8 weeks
  anxiety and depression Generalized Anxiety Disorder-7 Item Scale(GAD-7) and Patient Health Questionnaire-9 Scale (PHQ-9) assesses the possible presence of anxiety and depressive states. The GAD-7 and PHQ-9 is considered to be unbiased by the presence of somatic illness and is found to be reliable and valid . It consists of two sub-scales, anxiety and depression, both containing seven items.

SECONDARY OUTCOMES:
stigma | From enrollment to the end of treatment at 6 weeks
  The Social Impact Scale (SIS) was used to evaluate stigma associated with wound malodor. The SIS is widely used in patients with chronic diseases and includes 24 items within four dimensions, social exclusion, economic discrimination, inner sense of shame, and social isolation, evaluated using a Likert4 method. Total possible score ranged from 24 points to 96 points, with higher scores associated with a greater perceived social impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China